CLINICAL TRIAL: NCT05431894
Title: Behavioral and Recovery Support for 30 Day Post-Discharge Care in Participants With Cardiovascular Diseases
Brief Title: Behavioral and Recovery Support for 30 Day Post-Discharge Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laguna Health, Inc (Industry)
Collaborators: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EH21-092
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Cardiovascular Diseases
Keywords: Readmissions; Cardiovascular; Post-Discharge; Behavioral Health; Readmission Cost; 30 Day Readmission; Heart Failure; Care Management; Barriers to Care; Contextualizing Healthcare
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure

STUDY DESIGN:
Intervention Model Description: Participants were assigned upon consent randomly to an intervention or control group. The intervention group received support from Laguna Coaches for 30 days, the control group did not receive any support from Laguna coaches.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Group received support from Laguna Coaches
  Interventions: Behavioral: Laguna Coach Intervention Group
- Control Arm (No Intervention): Group received no support from Laguna Coaches

INTERVENTIONS:
Behavioral: Laguna Coach Intervention Group — Behavioral and mental support was delivered through personal interactions with Laguna Coaches via phone, video, or web chat. Behavioral and mental support was individualized to best match each patient's needs and strengths. Support was provided to participants through human interactions over approximately 30 days.
  Arms: Intervention Arm

SUMMARY:
This study will provide behavioral and mental health support to a select group of participants to supplement the hospital-provided discharge and recovery plans, based on clinical guidance and dedicated post-hospitalization behavioral protocols, with the goals of reducing readmission rates and costs.

DETAILED DESCRIPTION:
This study was designed to provide support to a select group of participants by supplementing the hospital-provided discharge instructions. Laguna integrated clinical guidance and dedicated post-hospitalization Laguna recovery protocols, with the aims of improving health outcomes, reducing health costs, and reducing readmission rates within 30 days post-discharge.

Participants in the intervention group received support from Laguna Health via phone, video, text, or web chat. Laguna provided contextual support to remove recovery barriers to these intervention participants.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the hospital with a diagnosis of a cardiovascular disease
* Discharged to home
* Converse in English or Spanish
* Uses a telephone

Exclusion Criteria:

* Participant unable to provide informed consent
* Participant lacks cognitive ability to participate in the study interventions as judged by the primary attending physician

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Unplanned All Cause Readmission Rate | 30 Days Post-Discharge
  Unplanned All-Cause 30 Day Readmission Rate
Unplanned Readmission Total Cost | 30 Days Post-Discharge
  Billed facility charges for readmissions hospitalization stays

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Tafur, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data

REFERENCES:
- [Background] Dieleman JL, Cao J, Chapin A, Chen C, Li Z, Liu A, Horst C, Kaldjian A, Matyasz T, Scott KW, Bui AL, Campbell M, Duber HC, Dunn AC, Flaxman AD, Fitzmaurice C, Naghavi M, Sadat N, Shieh P, Squires E, Yeung K, Murray CJL. US Health Care Spending by Payer and Health Condition, 1996-2016. JAMA. 2020 Mar 3;323(9):863-884. doi: 10.1001/jama.2020.0734. PMID 32125402
- [Background] Bailey MK, Weiss AJ, Barrett ML, Jiang HJ. Characteristics of 30-Day All-Cause Hospital Readmissions, 2010-2016. 2019 Feb 12. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #248. Available from http://www.ncbi.nlm.nih.gov/books/NBK538941/ PMID 30896914
- [Background] Panagiotou OA, Kumar A, Gutman R, Keohane LM, Rivera-Hernandez M, Rahman M, Gozalo PL, Mor V, Trivedi AN. Hospital Readmission Rates in Medicare Advantage and Traditional Medicare: A Retrospective Population-Based Analysis. Ann Intern Med. 2019 Jul 16;171(2):99-106. doi: 10.7326/M18-1795. Epub 2019 Jun 25. PMID 31234205
- [Background] Mitchell SE, Gardiner PM, Sadikova E, Martin JM, Jack BW, Hibbard JH, Paasche-Orlow MK. Patient activation and 30-day post-discharge hospital utilization. J Gen Intern Med. 2014 Feb;29(2):349-55. doi: 10.1007/s11606-013-2647-2. Epub 2013 Oct 4. PMID 24091935
- [Background] Riegel B, Masterson Creber R, Hill J, Chittams J, Hoke L. Effectiveness of Motivational Interviewing in Decreasing Hospital Readmission in Adults With Heart Failure and Multimorbidity. Clin Nurs Res. 2016 Aug;25(4):362-77. doi: 10.1177/1054773815623252. Epub 2016 Jan 6. PMID 26743119
- [Background] Villani A, Malfatto G, Compare A, Della Rosa F, Bellardita L, Branzi G, Molinari E, Parati G. Clinical and psychological telemonitoring and telecare of high risk heart failure patients. J Telemed Telecare. 2014 Dec;20(8):468-75. doi: 10.1177/1357633X14555644. Epub 2014 Oct 22. PMID 25339632
- [Background] Roncella A, Pristipino C, Cianfrocca C, Scorza S, Pasceri V, Pelliccia F, Denollet J, Pedersen SS, Speciale G. One-year results of the randomized, controlled, short-term psychotherapy in acute myocardial infarction (STEP-IN-AMI) trial. Int J Cardiol. 2013 Dec 10;170(2):132-9. doi: 10.1016/j.ijcard.2013.08.094. Epub 2013 Sep 8. PMID 24239154
- [Background] Allen LA, Smoyer Tomic KE, Smith DM, Wilson KL, Agodoa I. Rates and predictors of 30-day readmission among commercially insured and Medicaid-enrolled patients hospitalized with systolic heart failure. Circ Heart Fail. 2012 Nov;5(6):672-9. doi: 10.1161/CIRCHEARTFAILURE.112.967356. Epub 2012 Oct 16. PMID 23072736
- [Background] Bhalla R, Kalkut G. Could Medicare readmission policy exacerbate health care system inequity? Ann Intern Med. 2010 Jan 19;152(2):114-7. doi: 10.7326/0003-4819-152-2-201001190-00185. Epub 2009 Nov 30. PMID 19949133
- [Background] Ogunmoroti O, Osibogun O, Spatz ES, Okunrintemi V, Mathews L, Ndumele CE, Michos ED. A systematic review of the bidirectional relationship between depressive symptoms and cardiovascular health. Prev Med. 2022 Jan;154:106891. doi: 10.1016/j.ypmed.2021.106891. Epub 2021 Nov 17. PMID 34800472
- [Background] Levine GN, Cohen BE, Commodore-Mensah Y, Fleury J, Huffman JC, Khalid U, Labarthe DR, Lavretsky H, Michos ED, Spatz ES, Kubzansky LD. Psychological Health, Well-Being, and the Mind-Heart-Body Connection: A Scientific Statement From the American Heart Association. Circulation. 2021 Mar 9;143(10):e763-e783. doi: 10.1161/CIR.0000000000000947. Epub 2021 Jan 25. PMID 33486973
- [Background] Sreenivasan J, Abu-Haniyeh A, Hooda U, Khan MS, Aronow WS, Michos ED, Cooper HA, Panza JA. Rate, causes, and predictors of 90-day readmissions and the association with index hospitalization coronary revascularization following non-ST elevation myocardial infarction in the United States. Catheter Cardiovasc Interv. 2021 Jul 1;98(1):12-21. doi: 10.1002/ccd.29119. Epub 2020 Jul 20. PMID 32686892
- [Background] Reese RL, Freedland KE, Steinmeyer BC, Rich MW, Rackley JW, Carney RM. Depression and rehospitalization following acute myocardial infarction. Circ Cardiovasc Qual Outcomes. 2011 Nov 1;4(6):626-33. doi: 10.1161/CIRCOUTCOMES.111.961896. Epub 2011 Oct 18. PMID 22010201